CLINICAL TRIAL: NCT01469364
Title: Aztreonam Lysine for Inhalation (AZLI) in the Treatment of Early Bronchiolitis Obliterans Syndrome (BOS) After Lung Transplantation
Brief Title: Safety Study of Aztreonam Lysine for Inhalation (AZLI) in the Treatment of Early Bronchiolitis Obliterans Syndrome (BOS)
Acronym: AZLI
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00030559; Gilead Sciences, Inc (Other: Gileand Sciences, Inc); Pro00030191 (Other: Duke Site Protocol Number)
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Results first posted 2015-11-26 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2015-12

CONDITIONS: Complication of Transplanted Lung
Keywords: Lung Transplant; Lung Transplant Recipient
MeSH Terms: interventions — Inhalation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aztreonam Lysine for Inhalation (AZLI) (Experimental): Patients to received Aztreonam Lysine(AZLI)
  Interventions: Drug: Aztreonam Lysine for Inhalation (AZLI); Procedure: Status Post Lung Transplant

INTERVENTIONS:
Drug: Aztreonam Lysine for Inhalation (AZLI) — The intervention will involve open label treatment with AZLI inhaled 75mg TID self-administered intermittently for 28 days on study drug and 28 days off study drug over a study period of 5 consecutive months (on/off/on/off/on AZLI)
Procedure: Status Post Lung Transplant — Bronchoscopy, pulmonary function testing, and laboratory testing will be performed on a regular basis during study enrollment consistent with each center's usual standard clinical care.
  Other Names: Standard Post Lung Transplant Care

SUMMARY:
This study is a pilot two- center study to determine if aztreonam lysine for inhalation AZLI can be safely and self-administered in lung transplant recipients with newly diagnosed bronchiolitis obliterans syndrome, grade 1 (BOS) and obtain pilot data regarding its effect on lung function in order to appropriately design and power a larger multicenter randomized study.

The hypothesis is that AZLI is a safe and effective treatment for declining lung function in lung transplant recipients with early stage BOS.

DETAILED DESCRIPTION:
Lung transplantation is increasingly employed as a therapy for patients with advanced lung disease including cystic fibrosis, idiopathic pulmonary fibrosis or emphysema. Despite significant short-term improvements in life quality and measures of lung function after lung transplantation, long-term outcomes are disappointing primarily due to the development of a condition of airway fibrosis known as bronchiolitis obliterans (BO). It is hypothesized that aztreonam lysine for inhalation (AZLI) is a safe and effective treatment for declining lung function in lung transplant recipients with early stage BOS. In order to test the hypothesis, the investigators seek to establish the safety of AZLI in a two-center cohort of 30 lung transplant recipients with BOS treated intermittently for 5 consecutive study months and determine if this treatment leads to improvement or stabilization of lung function. The intervention will involve open label treatment with AZLI, in addition to usual transplant care, administered for 3 intermittent courses, 28 days each, over a 5 month study period.. Bronchoscopy, pulmonary function testing, and laboratory testing will be performed on a regular basis during study enrollment consistent with each center's usual standard clinical care. Patients will have a baseline screening visit, one month and five month study visit.. The study will take two years to complete from the start of funding. After a start-up period of 2 months, a total of 30 patients will be enrolled over 12 months across the two centers (15 patients each at DUMC and UCLA). Each enrolled patient will complete 5 months of intermittent therapy, and complete baseline, month 1 and month 5 visits. Over the next 6 months the study database will be finalized, statistical analysis will for primary and secondary outcomes will be performed leading to the generation of either a study abstract or manuscript.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 or older at the time of transplant) male or female
* Cadaveric first lung transplant recipient, single or bilateral; or multi-organ lung transplant recipient.
* Current FEV1 66-80% of posttransplant baseline FEV1, and meets all criteria for BOS 1 as defined by the International Society of Heart and Lung Transplantation.

  * Onset of BOS 1 within twelve months of screening

Exclusion Criteria:

* Known allergy to aztreonam
* Retransplant
* Pediatric patients
* Live lobar transplant recipients
* Inability to provide informed consent.
* Patients with advanced BOS (grades 2,3) or established BOS >6 months
* Pregnant Women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Palmer, MD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Belperio JA, Weigt SS, Fishbein MC, Lynch JP 3rd. Chronic lung allograft rejection: mechanisms and therapy. Proc Am Thorac Soc. 2009 Jan 15;6(1):108-21. doi: 10.1513/pats.200807-073GO. PMID 19131536
- [Background] Weigt SS, Wallace WD, Derhovanessian A, Saggar R, Saggar R, Lynch JP, Belperio JA. Chronic allograft rejection: epidemiology, diagnosis, pathogenesis, and treatment. Semin Respir Crit Care Med. 2010 Apr;31(2):189-207. doi: 10.1055/s-0030-1249116. Epub 2010 Mar 30. PMID 20354932
- [Background] Estenne M, Maurer JR, Boehler A, Egan JJ, Frost A, Hertz M, Mallory GB, Snell GI, Yousem S. Bronchiolitis obliterans syndrome 2001: an update of the diagnostic criteria. J Heart Lung Transplant. 2002 Mar;21(3):297-310. doi: 10.1016/s1053-2498(02)00398-4. No abstract available. PMID 11897517
- [Background] Lama VN, Murray S, Lonigro RJ, Toews GB, Chang A, Lau C, Flint A, Chan KM, Martinez FJ. Course of FEV(1) after onset of bronchiolitis obliterans syndrome in lung transplant recipients. Am J Respir Crit Care Med. 2007 Jun 1;175(11):1192-8. doi: 10.1164/rccm.200609-1344OC. Epub 2007 Mar 8. PMID 17347496
- [Background] Christie JD, Edwards LB, Kucheryavaya AY, Aurora P, Dobbels F, Kirk R, Rahmel AO, Stehlik J, Hertz MI. The Registry of the International Society for Heart and Lung Transplantation: twenty-seventh official adult lung and heart-lung transplant report--2010. J Heart Lung Transplant. 2010 Oct;29(10):1104-18. doi: 10.1016/j.healun.2010.08.004. No abstract available. PMID 20870165
- [Background] Finlen Copeland CA, Snyder LD, Zaas DW, Turbyfill WJ, Davis WA, Palmer SM. Survival after bronchiolitis obliterans syndrome among bilateral lung transplant recipients. Am J Respir Crit Care Med. 2010 Sep 15;182(6):784-9. doi: 10.1164/rccm.201002-0211OC. Epub 2010 May 27. PMID 20508211
- [Background] Vos R, Vanaudenaerde BM, Ottevaere A, Verleden SE, De Vleeschauwer SI, Willems-Widyastuti A, Wauters S, Van Raemdonck DE, Nawrot TS, Dupont LJ, Verleden GM. Long-term azithromycin therapy for bronchiolitis obliterans syndrome: divide and conquer? J Heart Lung Transplant. 2010 Dec;29(12):1358-68. doi: 10.1016/j.healun.2010.05.023. Epub 2010 Jul 8. PMID 20619683
- [Background] Gerhardt SG, McDyer JF, Girgis RE, Conte JV, Yang SC, Orens JB. Maintenance azithromycin therapy for bronchiolitis obliterans syndrome: results of a pilot study. Am J Respir Crit Care Med. 2003 Jul 1;168(1):121-5. doi: 10.1164/rccm.200212-1424BC. Epub 2003 Apr 2. PMID 12672648
- [Background] Vos R, Vanaudenaerde BM, Geudens N, Dupont LJ, Van Raemdonck DE, Verleden GM. Pseudomonal airway colonisation: risk factor for bronchiolitis obliterans syndrome after lung transplantation? Eur Respir J. 2008 May;31(5):1037-45. doi: 10.1183/09031936.00128607. Epub 2008 Feb 6. PMID 18256072
- [Background] Jain R, Hachem RR, Morrell MR, Trulock EP, Chakinala MM, Yusen RD, Huang HJ, Mohanakumar T, Patterson GA, Walter MJ. Azithromycin is associated with increased survival in lung transplant recipients with bronchiolitis obliterans syndrome. J Heart Lung Transplant. 2010 May;29(5):531-7. doi: 10.1016/j.healun.2009.12.003. Epub 2010 Feb 4. PMID 20133163
- [Background] McCoy KS, Quittner AL, Oermann CM, Gibson RL, Retsch-Bogart GZ, Montgomery AB. Inhaled aztreonam lysine for chronic airway Pseudomonas aeruginosa in cystic fibrosis. Am J Respir Crit Care Med. 2008 Nov 1;178(9):921-8. doi: 10.1164/rccm.200712-1804OC. Epub 2008 Jul 24. PMID 18658109
- [Background] Oermann CM, Retsch-Bogart GZ, Quittner AL, Gibson RL, McCoy KS, Montgomery AB, Cooper PJ. An 18-month study of the safety and efficacy of repeated courses of inhaled aztreonam lysine in cystic fibrosis. Pediatr Pulmonol. 2010 Nov;45(11):1121-34. doi: 10.1002/ppul.21301. PMID 20672296

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from two lung transplant centers, Duke and UCLA, and 30 subjects enrolled in the study from April 2013 to July 2014.
Period: Overall Study
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Started | 30
Completed | 28
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 30
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [33 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 28
  Black | 2
Region of Enrollment [Number; unit: participants]
  United States | 30
FEV1 [Median (Inter-Quartile Range); unit: liters] | 1.87 [1.57 to 2.46]
FVC [Median (Inter-Quartile Range); unit: liters] | 2.68 [2.34 to 3.22]
FEF 25-75 [Median (Inter-Quartile Range); unit: liters] | 1.18 [0.85 to 1.96]

OUTCOME MEASURES:

1. Primary Outcome: Change in Pulmonary Function, as Measured by Serial Forced Expiratory Volume in 1 Second (FEV1) on Spirometry
Description: Within-subject change to absolute FEV1 month 1 vs. 0. FEV1 was measured 14-35 days after the start of months 1 AZLI courses and compared to study month 0 (baseline/prior to 1st dose).
Time Frame: Baseline, month 1
Measure: Median (Inter-Quartile Range); unit: Liter
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 30
Liter | -0.04 [-0.22 to 0.12]
Statistical Analysis 1: Comparison: Aztreonam Lysine for Inhalation (AZLI); Test type: Superiority or Other; p = 0.2030, t-test, 2 sided; Paired t-test 2 sided

2. Primary Outcome: Change in Pulmonary Function, as Measured by Serial Forced Expiratory Volume in 1 Second (FEV1) on Spirometry
Description: Within-subject change to absolute FEV1 month 5 vs 0.
Time Frame: Baseline, month 5
Measure: Median (Inter-Quartile Range); unit: Liter
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 26
Liter | -0.02 [-0.25 to 0.10]
Statistical Analysis 1: Comparison: Aztreonam Lysine for Inhalation (AZLI); Test type: Superiority or Other; p = 0.2527, t-test, 2 sided; Paired t-test 2 sided

3. Secondary Outcome: Change in FEV1 Off AZLI Therapy
Description: This will be compared to study month 0 (baseline, when obtained as standard of care (SOC).
Time Frame: At Study Months 2 and 4
Population: Partial data for this outcome measure was collected on 4 participants and due to not having complete data set analyzation was not completed.
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in HRQOL Off AZLI Therapy.
Description: This will be compared to study month 0 (baseline), when obtained at standard of care visit (SOC)
Time Frame: At study months 2 or 4
Population: Partial data for this outcome measure was collected on 4 participants and due to not having a complete data set the analyzation was not completed.
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 0

5. Secondary Outcome: Among Patients Colonized With Pseudomonas Aeruginosa, Change in Infection Burden as Measured by the Culture Final Report (0,1+, 2+, 3+, 4+) of in Pseudomonas Aeruginosa Sputum or Bronchoalveolar Fluid.
Description: Microbiology data was collected when performed for SOC purposes on BAL or sputum samples. Baseline and 1 month value represents the culture final report value (0,1+, 2+, 3+, 4+) of Pseudomonas aeruginosa. A value of zero represents no Pseudomonas aeruginosa sputum or bronchoalveolar fluid. A value of 4 represents high amounts of Pseudomonas aeruginosa sputum or bronchoalveolar fluid.
Time Frame: Baseline, month 1
Population: The statistical analysis was unable to be performed due to insufficient number of paired observations. Only 9 of 30 enrolled had baseline microbiology data, 3 were cultured positive for Pseudomonas Aeruginosa. Only 1 of the 3 had a subsequent SOC BAL sample collected. Therefore, only raw data is entered for the one subject.
Measure: Number; unit: culture value of Pseudomonas aeruginosa
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 1
culture value of Pseudomonas aeruginosa
  Culture value at Baseline | 4
  Culture value at one month | 0

6. Secondary Outcome: Bronchoalveolar Lavage Fluid (BALF) Neutrophilia After Treatment, When Performed as Part of Clinical Care (SOC).
Description: The study team is measuring the change in neutrophils AFTER treatment. They will compare a SOC BAL taken after AZLI with the BAL taken within 90 days of AZLI initiation (pre or baseline measure). The post AZLI BAL measurement time range is 15 days after first course of AZLI up to last day of the 3rd and final course of AZLI (over a period of 5 consecutive months).
Time Frame: Baseline - defined as a within 90 days of enrollment and After Treatment (5 months)
Population: Participants with paired SOC bronchoalveolar lavage fluid cell differential counts performed within 90 days of AZLI month 1 (baseline timepoint) and >=15 days after AZLI dose 1 through the completion of dose 3 (study month 5) were included in the analysis (n=5).
Measure: Mean (Standard Deviation); unit: mean percentage of neutrophils
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 5
mean percentage of neutrophils | 7.80 (25.43)

7. Primary Outcome: Change in Global Health Related Quality of Life, Measured by Serially Self-administered Short Form 36 Health Survey Questionnaire (SF-36) at Baseline (Prior to AZLI First Dose) and During AZLI Therapy at Month 1
Description: The SF-36 is a commonly used, well validated measure of global health related quality of life. The survey was self-administered. There are 8 subscales which combine to form a Physical Component Score (PCS) and a Mental Component Score (MCS). We analyzed within subject changes to the PCS and MCS at month 1 vs. 0. MCS and PCS scores are relative to a US population mean of 50. The higher the score, the better one perceives his quality of life. A change in score of 4 points or more is considered clinically meaningful. Scores represent Median Absolute Difference. The SF-36 was completed 14-35 days after the start of months 1 AZLI courses and compared to study month 0 (baseline/prior to 1st dose).
Time Frame: Baseline, month 1
Population: subjects with completed SF-36 surveys at month 1 and month 0 (n=28)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 28
units on a scale
  PCS: month 1 vs. Baseline (n=28) | -1.52 [-4.21 to 2.71]
  MCS: month 1 vs. Baseline (n-28) | 0.78 [-0.96 to 5.42]
Statistical Analysis 1: Comparison: Aztreonam Lysine for Inhalation (AZLI); P-Value for the SF-36 PCS; Test type: Superiority or Other; p = 0.34, t-test, 2 sided; Paired Measured t-test; Mean Absolute Difference = -1.52
Statistical Analysis 2: Comparison: Aztreonam Lysine for Inhalation (AZLI); P-Value for the SF-36 MCS; Test type: Superiority or Other; p = 0.18, t-test, 2 sided; Paired Measured t-test; Median Absolute Difference = 0.78

8. Primary Outcome: Change in Global Health Related Quality of Life, Measured by Serially Self-administered Short Form 36 Health Survey Questionnaire (SF-36) at Baseline (Prior to AZLI First Dose) and During AZLI Therapy at Month 1 and Month 5.
Description: The SF-36 is a commonly used, well validated measure of global health related quality of life. The survey was self-administered. There are 8 subscales which combine to form a Physical Component Score (PCS) and a Mental Component Score (MCS). We analyzed within subject changes to the PCS and MCS at month 5 vs 0. MCS and PCS scores are relative to a US population mean of 50. The higher the score, the better one perceives his quality of life. A change in score of 4 points or more is considered clinically meaningful. Scores represent Median Absolute Difference. The SF-36 was completed 14-35 days after the start of months 1 and 5 AZLI courses and compared to study month 0 (baseline/prior to 1st dose).
Time Frame: Baseline, month 5
Population: subjects with completed SF-36 surveys at month 5 and 0 (n=26) time-points.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 26
units on a scale
  PCS: month 5 vs. Baseline (n=26) | 1.62 [-1.42 to 5.30]
  MCS: month 5 vs. Baseline (n-26) | -1.24 [-6.51 to 4.71]
Statistical Analysis 1: Comparison: Aztreonam Lysine for Inhalation (AZLI); P-Value for SF-36 PCS; Test type: Superiority or Other; p = 0.09, t-test, 2 sided; Paired Measure t-test; Median Absolute Difference = 1.62
Statistical Analysis 2: Comparison: Aztreonam Lysine for Inhalation (AZLI); P-Value for SF-36 MCS; Test type: Superiority or Other; p = 0.31, t-test, 2 sided; Paired Measure t-test; Median Absolute Difference = -1.24

9. Primary Outcome: Change in Respiratory-specific Health Related Quality of Life, Measured by Serially Self Administered St. George's Respiratory Questionnaire (SGRQ) at Baseline (Prior to AZLI First Dose) and During AZLI Therapy at Month 1
Description: The SRGQ measures activities, symptoms, and impacts of living with a pulmonary condition. We analyzed the change to the within-subject Total score month 1 vs. 0. Total score ranges from 0-100 with a smaller value representing better respiratory-specific QOL. A change in score of 4 points or more is considered clinically meaningful. Scores represent Median Absolute Difference in the Total Score. The SGRQ was completed 14-35 days after the start of months 1 AZLI courses and compared to study month 0 (baseline/prior to 1st dose).
Time Frame: Baseline, month 1
Population: subjects with completed SF-36 surveys at month 1 and month 0 (n=28) time-points.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 28
units on a scale | 0.82 [-6.53 to 8.20]
Statistical Analysis 1: Comparison: Aztreonam Lysine for Inhalation (AZLI); P-Value for SGRQ measure; Test type: Superiority or Other; p = 0.56, t-test, 2 sided; Paired Measure t-test; Median Absolute Difference = 0.82

10. Primary Outcome: Change in Respiratory-specific Health Related Quality of Life, Measured by Serially Self Administered St. George's Respiratory Questionnaire (SGRQ) at Baseline (Prior to AZLI First Dose) and During AZLI Therapy at Month 5.
Description: The SRGQ measures activities, symptoms, and impacts of living with a pulmonary condition. We analyzed the change to the within-subject Total score month 5 vs 0. Total score ranges from 0-100 with a smaller value representing better respiratory-specific QOL. A change in score of 4 points or more is considered clinically meaningful. Scores represent Median Absolute Difference in theTotal Score. The SGRQ was completed 14-35 days after the start of month 5 AZLI courses and compared to study month 0 (baseline/prior to 1st dose).
Time Frame: Baseline, month 5
Population: subjects with completed SF-36 surveys at month 5 and 0 (n=26) time-points.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 26
units on a scale | 0.15 [-5.21 to 6.19]
Statistical Analysis 1: Comparison: Aztreonam Lysine for Inhalation (AZLI); P-Value for SGRQ Measure; Test type: Superiority or Other; p = 0.68, t-test, 2 sided; Paired Measure t-test; Median Absolute Difference = 0.15

11. Primary Outcome: Change in Pulmonary Function, as Measured by Serial Forced Expiratory Flow (FEF25-75) on Spirometry at Baseline (Prior to AZLI First Dose) and During AZLI Therapy at Month 5.
Description: Within-subject change to absolute FEF 25-75 month 5 vs 0. FEF 25-75 was measured 14-35 days after the start of months 5
Time Frame: Baseline, month 5
Measure: Median (Inter-Quartile Range); unit: Liter
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 26
Liter | -0.015 [-0.360 to 0.170]
Statistical Analysis 1: Comparison: Aztreonam Lysine for Inhalation (AZLI); Test type: Superiority or Other; p = 0.7454, t-test, 2 sided; Paired t-test 2 sided

12. Primary Outcome: Change in Pulmonary Function, as Measured by Serial Forced Expiratory Flow (FEF25-75) on Spirometry at Baseline (Prior to AZLI First Dose) and During AZLI Therapy at Month 1
Description: Within-subject change to absolute FEF 25-75 month 1 vs. 0. FEF 25-75 was measured 14-35 days after the start of months 1
Time Frame: Baseline, month 1
Measure: Median (Inter-Quartile Range); unit: Liter
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Number analyzed (Participants) | 30
Liter | -0.025 [-0.190 to 0.130]
Statistical Analysis 1: Comparison: Aztreonam Lysine for Inhalation (AZLI); Test type: Superiority or Other; p = 0.9638, t-test, 2 sided; Paired t-test was completed

ADVERSE EVENTS:
Time Frame: Adverse events were collected on study day 1, day 7 and at the end of study month 1 and 5.
Arm/Group | Aztreonam Lysine for Inhalation (AZLI)
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 13/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aztreonam Lysine for Inhalation (AZLI) (N=30)
Left pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aztreonam Lysine for Inhalation (AZLI) (N=30)
Cough during or after administration (Respiratory, thoracic and mediastinal disorders) | 13
Dry mouth during administration (General disorders) | 2
Increased dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Increased sputum production (Respiratory, thoracic and mediastinal disorders) | 2
Thinned out mucous (Reproductive system and breast disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dysphonia (General disorders) | 1
Irritability (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No